CLINICAL TRIAL: NCT07163546
Title: Investigation of the Outcomes of the Person-Centered Lifestyle Redesign in Individuals With Chronic Low Back Pain
Brief Title: Person-Centered Lifestyle Redesign in Chronic Low Back Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Etkin Bagi, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-ERG-EB-02
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain, Chronic
Keywords: pain; quality of life; disability; physical activity; mental status; occupational therapy
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention and Physical therapy (Experimental): It is a group that receives physical therapy and lifestyle intervention.
  Interventions: Behavioral: Lifestyle intervention
- Physical therapy (No Intervention): This group only receives physical therapy

INTERVENTIONS:
Behavioral: Lifestyle intervention — A lifestyle intervention is an occupational therapy intervention program that aims to help individuals change their lifestyle by encouraging greater engagement in meaningful activities. This program aims to help participants develop healthy routines and habits. It offers a perspective that combines various approaches such as patient education, occupational self-analysis, problem-solving, and building motivation to prevent and manage chronic health problems. Participants gain self-analysis and problem-solving skills while experiencing positive lifestyle changes and developing healthy routines.
  The lifestyle intervention was planned as a total of 8 sessions, 2 sessions per week.
  Arms: Lifestyle intervention and Physical therapy

SUMMARY:
This study is designed to examine the effects of a person-centered lifestyle intervention on pain, occupational performance, quality of life, disability, physical activity levels, and mental status in individuals with chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is the most common musculoskeletal disorder worldwide; 70-80% of the adult population experiences this condition at some point in their lives. It is considered a leading cause of workforce loss and years lived with functional disability, and it ranks among the top five most frequent diagnoses in primary healthcare. Chronic low back pain is a significant public health problem globally, associated with substantial discomfort, disability, medical costs, and economic burden.

Chronic low back pain can severely reduce quality of life and has a significant comorbidity with mental health; therefore, it not only restricts an individual's physical activities and daily tasks but also negatively impacts psychological well-being, leading to higher levels of subclinical depression and anxiety. Non-surgical treatment options for chronic low back pain include pharmacological and non-pharmacological therapies.

Within the pharmacological approach, non-steroidal anti-inflammatory drugs (NSAIDs) and opioids are commonly prescribed. Despite their therapeutic efficacy, this approach has significant drawbacks. It provides limited improvement in pain and functional limitations for most patients, which is frustrating. Furthermore, the long-term use of NSAIDs and opioids can cause serious side effects such as gastrointestinal bleeding, arterial thrombosis, addiction, and mental dysfunction.

While non-pharmacological therapies individually have positive effects, there is a lack of conclusive evidence supporting the superiority of one approach over others. Consequently, the treatment process should be tailored to the needs of the individual with chronic low back pain, and it appears that combined therapies addressing the individual holistically are needed to achieve effective results. The biopsychosocial approach to treating chronic pain considers biological, psychological, and social factors. Clinical guidelines for chronic low back pain have shown a shift towards the biopsychosocial model. This can provide clinicians with some insights into additional areas to consider in their patients' treatment.

Lifestyle risk factors such as excess weight, physical inactivity, poor nutrition, and smoking play a role in the development of low back pain. Studies suggest that addressing such lifestyle factors can improve outcomes in low back pain, including disability. Despite evidence suggesting the potential benefits of interventions targeting these lifestyle factors, only one randomized controlled trial has been conducted for patients with chronic low back pain. This study found no effect, largely due to insufficient adherence to the treatment.

A lifestyle intervention is an occupational therapy intervention program that aims to help individuals change their lifestyle by encouraging greater engagement in meaningful activities. This program aims to help participants develop healthy routines and habits. It offers a perspective that combines various approaches such as patient education, occupational self-analysis, problem-solving, and building motivation to prevent and manage chronic health problems. Participants gain self-analysis and problem-solving skills while experiencing positive lifestyle changes and developing healthy routines.

Our study was planned to investigate the effects of a person-centered lifestyle intervention on pain, occupational performance, quality of life, disability, physical activity levels, and mental status in individuals with chronic low back pain, due to the limited number of studies conducted on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years old
* Lower back pain lasting ≥3 months
* Pain at least 4 according to VAS
* Being literate

Exclusion Criteria:

* Presence of congenital or acquired spinal deformity (scoliosis, kyphosis, spondylolisthesis),
* Presence of history of spinal surgery (<12 months) (spinal fusion, discectomy),
* Diagnosis of radiculopathy or neuropathy (spinal canal stenosis),
* Presence of serious fractures or pathologies (vertebral fractures, infections),
* Presence of malignancy,
* Presence of chronic cardiovascular and pulmonary diseases,
* Severe psychiatric, neurological, infectious, renal or inflammatory disorders,
* Systematic metabolic disorder,
* Pregnancy
* BMI ≥ 30 kg/m²

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | six months
  The Visual Analog Scale (VAS) is a simple, effective, valid, and reliable tool that is internationally recognized for assessing participants' pain intensity. Participants are asked to mark on a 10 cm horizontal line to indicate how severely they perceive their pain. The left end of the scale represents "no pain" (0 cm), and the right end represents "unbearable pain" (10 cm). Assessment is performed by precisely measuring the horizontal distance of the marked point from the left end with a ruler. This numerical value is interpreted as an indicator of the participant's pain severity. A score between 1-3.9 cm indicates mild pain, 4-6.9 cm indicates moderate pain, and 7-10 cm indicates severe pain.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | six months
  The COPM is a semi-structured assessment tool that allows individuals to identify performance areas in daily life where they experience problems and to measure their level of occupational performance and satisfaction in these areas. It consists of three sections: self-care, leisure, and productivity. In the first stage, the individual is asked to rate the importance of their activities in these three areas on a scale of 1 to 10 (1: not important at all, 10: extremely important). In the next stage, the individual selects the five activities they identified as most important. For each selected activity, they are asked to rate both their performance (1: my performance is very poor, 10: my performance is very good) and their satisfaction (1: not satisfied at all, 10: extremely satisfied) on a Likert-type scale from 1 to 10. For scoring, the performance scores given for each activity are summed and divided by the number of selected activities to obtain an average
Nottingham Health Profile (NHP) | six months
  The Nottingham Health Profile subjectively evaluates an individual's health status through 38 items across six different dimensions: emotional reactions (9 items), physical mobility (8 items), pain (8 items), sleep (5 items), social isolation (5 items), and energy level (3 items). Participants are required to answer the questions with 'yes' or 'no'. The score for each sub-dimension is calculated on a scale from 0 to 100, and the maximum total score obtained by summing all dimension scores is 600. In the interpretation of the scores, a lower total score is associated with a better quality of life. The reported Cronbach's alpha values for the different sub-dimensions of the scale range from 0.56 to 0.83.
Oswestry Disability Index (ODI) | six months
  The Oswestry Disability Index examines 10 different dimensions affecting daily life: pain intensity, personal care, lifting, walking, sitting, standing, sleep quality, sex life, social life, and traveling. The lowest possible score on the scale is 0, and the highest is 50. The total score is multiplied by 2 to express the individual's disability level as a percentage (%). An increase in the score indicates an increase in the level of disability experienced by the individual due to low back pain. The Cronbach's alpha value of the ODI is 0.89, stating that the scale is highly reliable.
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | six months
  The International Physical Activity Questionnaire - Short Form is to objectively assess individuals' physical activity levels over the last seven days. Consisting of four sections and seven questions, the questionnaire asks the participant to recall and report physical activities performed for at least 10 minutes at a time during the last seven days. The questionnaire collects information on the time spent walking, in moderate-intensity activities, and in vigorous-intensity activities, as well as sedentary time spent sitting. These duration data are converted into a Metabolic Equivalent (MET)-minute/week score to express physical activity in terms of energy expenditure. Standard, internationally accepted MET values are used for this calculation: Walking: 3.3 METs, Moderate Physical Activity: 4.0 METs, Vigorous Physical Activity: 8.0 METs, Sitting: 1.5 METs.
Hospital Anxiety and Depression Scale (HADS) | six months
  The Hospital Anxiety and Depression Scale is to screen participants' anxiety and depression levels. The scale consists of 14 items total and comprises two subscales: Anxiety (HADS-A) and Depression (HADS-D), each containing 7 items. Participants are asked to respond to each item on a four-point Likert-type scale ranging from 0 to 3. The score for each subscale ranges from 0 to 21. Higher scores indicate greater severity of symptoms in the respective dimension. The Cronbach's alpha coefficients for the scale were reported as 0.85 for anxiety and 0.77 for depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No